CLINICAL TRIAL: NCT02787031
Title: Sources of Variation in Anesthesia Care for Hip Fracture Surgery and the Association With Outcomes
Brief Title: Variations in Anesthesia Care for Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM2
Record Dates: First submitted 2016-05-17; First posted 2016-06-01 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Hip Fractures; Anesthesia; Death
Keywords: hip fracture; geriatric; epidemiology; practice variation; anesthesia
MeSH Terms: conditions — Hip Fractures; Death | interventions — Anesthesia, Spinal; Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neuraxial anesthesia: Participants in this group will be those who had a spinal or epidural anesthetic without concurrent general anesthesia
  Interventions: Procedure: Neuraxial anesthesia
- General anesthesia: Participants in this group will be those who had general anesthesia, including those who had a general plus a concurrent spinal or epidural anesthetic.
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Neuraxial anesthesia
  Other Names: spinal anesthesia; epidural anesthesia
  Groups: Neuraxial anesthesia
Procedure: General anesthesia
  Groups: General anesthesia

SUMMARY:
The investigators will use health administrative data to examine the variation of anesthesia type for hip fracture surgery, as well as sources of variation and predictors of variation.

DETAILED DESCRIPTION:
To evaluate the sources of variance in utilization of neuraxial anesthesia the investigators will use multilevel multivariable modeling strategies. This will allow identification of sources of variation (hospital, vs physician, vs patient characteristics), as well as identification of independent predictors of neuraxial use at each of these three levels.

The investigators will also evaluate the independent association of hospital level variation in neuraxial use on our outcomes of interest using multilevel multivariable regression.

ELIGIBILITY:
Inclusion Criteria:

* Had hip fracture surgery
* Admitted to hospital on a non-elective basis

Exclusion Criteria:

* Do not hold a valid provincial health insurance account

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All Ontario residents aged 66 years or older on the day of their emergency hip fracture surgery.
Sampling Method: Non-Probability Sample
Enrollment: 107317 (Actual)
Dates: Start 2002-04; Primary Completion 2013-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McIsaac, MD,MPH,FRCPC, Principal Investigator — The Ottawa Hospital
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McIsaac DI, Wijeysundera DN, Bryson GL, Huang A, McCartney CJL, van Walraven C. Hospital-, Anesthesiologist-, and Patient-level Variation in Primary Anesthesia Type for Hip Fracture Surgery: A Population-based Cross-sectional Analysis. Anesthesiology. 2018 Dec;129(6):1121-1131. doi: 10.1097/ALN.0000000000002453. PMID 30273269

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuraxial Anesthesia: Participants in this group will be those who had a spinal or epidural anesthetic without concurrent general anesthesia
  Neuraxial anesthesia
- General Anesthesia: Participants in this group will be those who had general anesthesia, including those who had a general plus a concurrent spinal or epidural anesthetic.
  General anesthesia
Period: Overall Study
Arm/Group | Neuraxial Anesthesia | General Anesthesia
Started | 57080 | 50237
Completed | 57080 | 50237
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuraxial Anesthesia | General Anesthesia | Total
Number analyzed (Participants) | 57080 | 50237 | 107317
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (7) | 82 (8) | 83 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41954 | 36874 | 78828
  Male | 15126 | 13363 | 28489
Neighbourhood income quintile [Median (Inter-Quartile Range); unit: Neighbourhood income quintile] — Neighborhood socioeconomic status of the participants is presented as income quintile (income quintile is a measure of neighbourhood socioeconomic status that divides the population into five income groups (from lowest income to highest income)). The scale is from 1-5 (income group quintile 1 (lowest), 2, 3, 4, 5 (highest)).
  Neighbourhood income quintile | 3 [2 to 4] | 3 [2 to 4] | 3 [2 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Cause Mortality at 30-days
Time Frame: Day of surgery to day of death, or up to 30 days, whichever comes first
Population: Data were not collected from the participants in the "General Anesthesia" Arm/Group. Only neuraxial group data available for all cause 30-day mortality. The aim was to measure the association of hospital-level utilization of neuraxial anesthesia, independent of patient-level use, with 30-day survival and length of stay and costs.
Measure: Count of Participants; unit: Participants
Arm/Group | Neuraxial Anesthesia | General Anesthesia
Number analyzed (Participants) | 57080 | 0
Participants | 9122 |

2. Secondary Outcome: Healthcare Costs From the Perspective of the Universal Healthcare System, Using Standardized Methods (Health System Performance Research Network 2013)
Time Frame: Day of surgery to day of death, or 30 days after surgery, whichever comes first
Population: Data were not collected from the participants in the "General Anesthesia" Arm/Group. Only neuraxial group data available for healthcare costs. The aim was to measure the association of hospital-level utilization of neuraxial anesthesia, independent of patient-level use, with 30-day survival and length of stay and costs.
Measure: Median (Inter-Quartile Range); unit: Canadian Dollars
Arm/Group | Neuraxial Anesthesia | General Anesthesia
Number analyzed (Participants) | 57080 | 0
Canadian Dollars | 22138 [16430 to 28354] |

3. Other Pre Specified Outcome: Hospital Length of Stay
Time Frame: Day of surgery to day of discharge, or up to 365 days, whichever comes first
Population: Data were not collected from the participants in the "General Anesthesia" Arm/Group. Only neuraxial group data available for hospital length of stay The aim was to measure the association of hospital-level utilization of neuraxial anesthesia, independent of patient-level use, with 30-day survival and length of stay and costs.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Neuraxial Anesthesia | General Anesthesia
Number analyzed (Participants) | 57080 | 0
Days | 9 [6 to 18] |

ADVERSE EVENTS:
Time Frame: 30 Days
Description: All-Cause Mortality: The occurrence of death due to any cause was reported. No other AEs were collected or monitored.
Arm/Group | Neuraxial Anesthesia | General Anesthesia
All-Cause Mortality (participants affected / at risk) | 9122/57080 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Health administrative data are not initially collected for research purposes. There are patient-level predictors, hospital-level variables, and anesthesiologist variables that we could not measure directly. Surgeon-specific variables such as preference for neuraxial versus general anesthesia could influence anesthesia decision making and should be considered. Patient-preference should contribute to warranted variation. The generalizability of our findings to other jurisdictions is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No